CLINICAL TRIAL: NCT03064776
Title: Pilot Study of m-RESIST, an m-Health Program for Treatment-resistant Schizophrenia: Acceptability, Usability, Satisfaction and Perceived Quality of Life Reported by Patients and Caregivers
Brief Title: Study of m-RESIST, an m-Health Program for Treatment-resistant Schizophrenia
Acronym: m-RESIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Sheba Medical Center (Other Government); Semmelweis University (Other); iMinds (Industry); AQuAS, Agència de Qualitat i Avaluació Sanitàries (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-RES-2016-51; 643552 (Other Grant/Funding Number: EU Horizon2020 research & innovation programme)
Record Dates: First submitted 2016-10-17; First posted 2017-02-27 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2019-06

CONDITIONS: Schizophrenia
Keywords: telemedicine
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- m-RESIST Patients (Experimental): m-RESIST is a system designed to improve illness self-management and facilitate recovery in individuals with Treatment-resistant schizophrenia (TRS). The system will be used to
  1. Continuously capture multidimensional behaviour as it occurs in real-time and in real-world environments, using continuous collection and analysis of sensor data.
  2. Detect individual early warning signs, and trigger targeted interventions that may mitigate the severity of worsening or prevent their recurrence altogether, using the clinical decision support system (CDSS) and Recommender operation.
  The m-RESIST will deliver both system initiated (i.e. pre-programmed) and patient-initiated (i.e. on-demand) real-time assessments, to the participants and in their own environment.
  Interventions: Device: m-RESIST Patients
- m-RESIST Caregivers (Experimental): m-RESIST is a system designed to improve illness self-knowledge and facilitate the involvement of caregivers in treatment of individuals with treatment-resistant schizophrenia.
  Interventions: Device: m-RESIST Caregivers

INTERVENTIONS:
Device: m-RESIST Patients — A mobile system based on Information and Communications Technology (ICT), which is addressed to empower patients suffering from TRS and to involve their caregivers
  Arms: m-RESIST Patients
Device: m-RESIST Caregivers — A mobile system based on Information and Communications Technology (ICT), which is addressed to empower patients suffering from TRS and to involve their caregivers
  Arms: m-RESIST Caregivers

SUMMARY:
m-RESIST is an m-health intervention program aimed to develop, test and evaluate a tool to allow patients suffering from treatment-resistant schizophrenia to self-manage their condition. This may facilitate acceptance and involvement of patients with their own treatment, as well as of caregivers. Moreover this programme could provide a new tool to the psychiatrist, psychologists working together with other health care professionals, to better monitor patients, through a personalised and optimised therapeutic process.

The present document corresponds to the pilot field-trials phase included in a three year European research project, co-funded by the Horizon 2020 Framework Programme of the European Union (grant agreement nº 643552). This document summarises the protocol of the whole therapeutic process, specifying all the procedures included in the program. This protocol will be implemented in three countries: Israel, Hungary and Spain, in order to test acceptability, usability, satisfaction and changes in the quality of life reported by the end-users.

DETAILED DESCRIPTION:
The main goal of the present study is to evaluate the acceptability, usability, and satisfaction to m-RESIST solution among the target groups (patients, caregivers, clinicians), and also to evaluate the effect of m-RESIST solution to empowerment and perceived quality of life of the treatment-resistant Schizophrenia patients (TRS). Interventions targeting key problems in TRS (risk behaviours, persistent symptoms of psychosis, poor medication adherence, unhealthy lifestyle habits) will be administered in a clinical setting, with the long-term goal of creating a widely-available system that can be deployed by users as needed, in their own environments.

The study will be conducted in three different regions: Gertner (Israel), Semmelweis (Hungary) and Barcelona (Spain). Consequently, the outcomes obtained in each site and their comparison will allow improving the m-RESIST program in terms of interoperability, integration of components and final implementation of the interactive system in the healthcare pathways.

The participants will be selected from Sheba Medical Center - Psychiatric Division (Tel Aviv), Semmelweis University - Department of Psychiatry and Psychotherapy (Budapest), and the adult psychiatric outpatient service of Hospital de la Santa Creu i Sant Pau (Barcelona).

A total of 45 patients with TRS (15 per centre), with their caregiver, will be included in the trial. All participants will be fully informed about the nature of the study (aims, methodology) and the system tested (data protection, expected risks/benefits, possible adverse events) and they will sign the informed consent for their participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Schizophrenia following the diagnostic and statistical manual of mental disorders (DSM-V) criteria.
* Meet criteria for "treatment-resistant schizophrenia", term referred to two different subgroups of patients:

  * Patients with schizophrenia who are refractory despite receiving antipsychotic treatment in suitable doses and duration (at least two dopamine D2 receptors antagonist antipsychotics, or on-going treatment with clozapine due to meeting treatment-resistant criteria), and presenting good adherence to treatment (Peuskens, 1999).
  * Patients who may be considered pseudo-resistant to the treatment or resistance-like (Elkis & Meltzer, 2007). In this case, presence of active symptoms may be influenced by psychiatric and medical conditions such as poor insight, negative attitude to medication, social isolation, consumption of toxic substances, presence of nutritional and medical problems, inappropriate health habits, as well as poor alliance and/or environment conditions (low involvement of caregivers in the therapeutic process), which may substantially contribute to poor responses or insufficient effects of medication.
* Duration of disease less than 15 years.
* Used to Information and Communication Technologies (ICT) and having the physical capability to use them (determined using the Technological Readiness Questionnaire).
* Presence of a informal caregiver -family members or significant others- of patients with treatment-resistant schizophrenia.

Exclusion Criteria:

* Meet criteria for remission according to the Remission of Schizophrenia Working Group (Andreasen et al., 2005.)
* The presence of delusions mainly related with their therapists or with new technologies.
* Hearing, vision, or motor impairment that makes it impossible to operate a smartphone.
* Presence of a caregiver or Informal carer not used to ICT or physical incapability to use them (determined using the Technological Readiness Questionnaire).
* Presence of intellectual developmental disability.-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Technology Acceptance Model (TAM) | Changes from baseline scores at 1-month and 3-months scores

SECONDARY OUTCOMES:
Change in User Experience Questionnaire | Changes from baseline scores at 1-month and 3-months scores
Change in EuroQol-5D Health Questionnaire (EQ-5D) | Changes from baseline scores at 1-month and 3-months scores
Change in Client Satisfaction Questionnaire (CSQ-8) | Changes from baseline scores at 1-month and 3-months scores
Change in Positive and Negative Syndrome Scale for Schizophrenia (PANSS) | Changes from baseline scores at 1-month and 3-months scores
Change in Neuropsychological Assessment | Changes from baseline scores at 1-month and 3-months scores
Change in Clinical Global Impression-Schizophrenia (CGI-SCH) | Changes from baseline scores at 1-month and 3-months scores
Change in Social Functioning Scale (SFS) | Changes from baseline scores at 1-month and 3-months scores

CONTACTS AND LOCATIONS:
Overall Officials: Corripio Iluminada, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (3):
- 3Department of Psychiatry and Psychotherapy, Semmelweis University, Budapest, Hungary
- The Gertner Institute of Epidemiology and Health Policy Research, Sheba Medical Center, Tel Aviv, Israel
- Department of Psychiatry. Hospital Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grasa E, Seppala J, Alonso-Solis A, Haapea M, Isohanni M, Miettunen J, Caro Mendivelso J, Almazan C, Rubinstein K, Caspi A, Unoka Z, Farkas K, Usall J, Ochoa S, van der Graaf S, Jewell C, Triantafillou A, Stevens M, Reixach E, Berdun J; m-RESIST group; Corripio I. m-RESIST, a Mobile Therapeutic Intervention for Treatment-Resistant Schizophrenia: Feasibility, Acceptability, and Usability Study. JMIR Form Res. 2023 Jun 30;7:e46179. doi: 10.2196/46179. PMID 37389933
- [Derived] Alonso-Solis A, Rubinstein K, Corripio I, Jaaskelainen E, Seppala A, Vella VA, Caro-Mendivelso J, Caspi A, Isohanni M, Unoka Z, Van der Graff S, Farkas K, Huerta-Ramos E, Marco-Garcia S, Stevens M, Coenen T, Hospedales M, Berdun J; m-Resist group; Grasa EM. Mobile therapeutic attention for treatment-resistant schizophrenia (m-RESIST): a prospective multicentre feasibility study protocol in patients and their caregivers. BMJ Open. 2018 Jul 16;8(7):e021346. doi: 10.1136/bmjopen-2017-021346. PMID 30012788